CLINICAL TRIAL: NCT04410393
Title: Comparison of the Sacrocolpopexy Operation and Lateral Suspension Operations Performed in the Treatment of Vaginal Cuff Prolapse in Patients With Hysterectomized Patients
Brief Title: Sacrocolpopexy and Lateral Suspension Operations
Status: Active, not recruiting | Type: Observational
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Pınar Kadirogulları, Pınar Kadiroğulları M.D, Department of Obstetrics and Gynecology,Principal Investigator, Kanuni Sultan Suleyman Training and Research Hospital
Other Study IDs: ATADEK- 2020/06
Record Dates: First submitted 2020-05-27; First posted 2020-06-01 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-07

CONDITIONS: Prolapse; Cuff
Keywords: sacrocolpopexy; Lateral Suspension
MeSH Terms: conditions — Prolapse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- sacrocolpopexy patients: Patients who underwent sacrocolpopexy for the treatment of vaginal cuff prolapse in patients who had previously undergone hysterectomy for benign causes
  Interventions: Procedure: vaginal cuff prolapse surgery
- lateral suspension surgery patients: Patients who underwent lateral suspension surgery for vaginal cuff prolapse in patients who had previously undergone hysterectomy for benign causes
  Interventions: Procedure: vaginal cuff prolapse surgery

INTERVENTIONS:
Procedure: vaginal cuff prolapse surgery — Different surgical methods for the treatment of vaginal cuff prolapse in patients who have previously undergone hysterectomy for benign causes

SUMMARY:
Different surgical methods can be used in the treatment of vaginal cuff prolapse in patients who had previously undergone hysterectomy for benign reasons. One of these is sacrocolpopexy and the other is lateral suspension. the investigators want to compare the results of patients undergoing these two operations. Thus, the difference between surgical methods will be investigated.

DETAILED DESCRIPTION:
Patients with symptomatic vaginal cuff prolapse will be operated; There will be two kinds of operation. After the operations, the patients will be followed up, a questionnaire will be applied to the postoperative patients and some questions will be asked. Pelvic examinations will also be performed and they will be evaluated for recurrence and complication. At the end of the study, the data of both groups will be compared and their superiority to each other will be shown.

ELIGIBILITY:
Inclusion Criteria:

* Patients who had previously undergone hysterectomy for benign causes
* Patients with symptomatic vaginal cuff prolapse during hysterectomy follow-up
* And for this, patients scheduled for operation

Exclusion Criteria:

* Patients with chronic diseases or medications that interfere with the operation
* Patients with oncology operated for malignant cause
* Non-localized patients with vaginal cuff prolapse

Ages: 40 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Different surgical methods can be used in the treatment of vaginal cuff prolapse in patients who had previously undergone hysterectomy for benign reasons. One of these is sacrocolpopexy and the other is lateral suspension. The investigators will form study groups of patients who underwent these two operations.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
recurrence | 1 years
  Patients will be followed up for 1 year after surgery and will be evaluated for recurrence at 1, 6 and 12 months.
  degree of uterine desensus cystocele and rectocele degree to be examined Recurrence rate will be defined by pelvic examination according to POP-Q scoring.
complications | 1 years
  Patients will be followed up for 1 year after the operation and will be evaluated for complications at 1, 6 and 12 months.
  bleeding ( bleeding rate will be specified in milliliters ) the risk of infection (According to the findings, there is an infection with / without infection.)

CONTACTS AND LOCATIONS:
Locations (1):
- Kanuni Sultan Süleyman Training and Research Hospital, Istanbul, Turkey (Türkiye)